CLINICAL TRIAL: NCT00245271
Title: Double-Blind, Multicenter Study Evaluating the Safety of OMS103HP and Vehicle in Subjects Undergoing Anterior Cruciate Ligament Reconstruction With an Open-Label Phase Containing a PK Analysis in a Subset of Subjects
Brief Title: Safety of OMS103HP in Patients Undergoing Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Gregory Demopulos, MD, CEO, CMO, Omeros Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C04516
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Knee; Musculoskeletal System; Ligament; ACL reconstruction
MeSH Terms: interventions — OMS 103HP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): OMS103 Irrigation Solution
  Interventions: Drug: OMS103HP
- 2 (Placebo Comparator): Balanced Salt Solution (BSS)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS103HP — Maximum of 13 bags of OMS103HP irrigation solution over a maximum of 2 hours
  Arms: 1
Drug: Vehicle — Maximum of 13 bags of BSS irrigation over a maximum of 2 hours.
  Arms: 2

SUMMARY:
OMS103HP is being developed for improvement in knee function following ACL reconstruction. Secondary benefits being evaluated include reduced postoperative pain, improvement in knee motion and earlier return to work.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) is an important stabilizer of the knee. Orthopedic surgeons replace the torn ligament during ACL reconstruction surgery. Surgical trauma initiates an acute inflammatory response, including swelling and pain, that leads to restricted joint motion and loss of function. Because of the dynamic nature, complexity and redundancy of the chemical mediators of inflammation and pain and their pathways, no currently available single drug has sufficiently broad spectrum of activity to effectively inhibit the inflammatory process. OMS103 provides a multicomponent approach to controlling the inflammation induced by arthroscopic surgery. It delivers three active ingredients, each with distinct pharmacological activities, directly to the site of surgical procedures to preemptively block the inflammatory cascade induced by surgical trauma.

ELIGIBILITY:
Inclusion Criteria:

* 17 - 65 years of age
* In good general health
* Undergoing arthroscopic ACL reconstruction for an ACL tear

Exclusion Criteria:

* Allergies to any of the individual ingredients in OMS103HP
* Has open physes in the distal femur or proximal tibia
* Undergoing bilateral knee surgery
* Subject who is considered by Investigator to be an unsuitable candidate

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2004-10; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The overall incidence of adverse events regardless of relationship to study drug. | 90 days

SECONDARY OUTCOMES:
Measures of safety and tolerability (e.g., clinical laboratory tests, physical examinations, etc.). | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Omeros Corporation
Locations (10):
- United States (10):
  - Kerlan-Jobe Orthopaedic Clinic, Los Angeles, California
  - Sports, Orthopedic and Rehabilitation Medicine Associates (S.O.A.R.), Redwood City, California
  - Advanced Orthopedic and Sports Medicine Specialists, Denver, Colorado
  - Colorado Orthopedic Consultants, PC, Englewood, Colorado
  - Rush University, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Sports Medicine, Columbus, Ohio
  - Temple University Orthopedics, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania